CLINICAL TRIAL: NCT00314613
Title: Functional Brain Imaging and Employment in First-Episode Psychotic Patients Treated With Risperdal
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Janssen, LP (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 7858; 7858; RIS-NAP-4007
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2010-05

CONDITIONS: Schizophrenia
Keywords: Schizophreniform; Schizophrenia; Schizoaffective Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Antipsychotic Agents

INTERVENTIONS:
Drug: Antipsychotic/Risperidone Consta

SUMMARY:
Assured treatment with Risperal CONSTA will provide first-episode patients, who have a greater potential for therapeutic response, with their best opportunity for continued improvement in cognitive function beyond three months of treatment.

DETAILED DESCRIPTION:
First episode patients have a greater potential for therapeutic response than multi-episode patients, and many of them also havea great desire to rejoin the workforce. Unfortunately, first episode patients become non-compliant or intermittently compliant with prescribed antipsychotic treatment at least as frequently as multi-episode patients. We believe that assured treatment with Risperal CONTSTA will provide first episode patients wiwth their best opporutnity for continued improvement in cognitive function beyond 3 months of treatment and that improvements in cognitive function will be associated with a greater likelihood of employment, real-world outcomes, such as independent living, as well as measures of brain function.

ELIGIBILITY:
Inclusion Criteria:

* male or female between 18-40 years of age
* meet DSM-IV criteria for first-episode schizophreniform, schizophrenia or schizoaffective disorder

Exclusion Criteria:

* pregnant & breast-feeding women
* patients with known sensitivity to oral Risperdal

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William H Wilson, PhD, Principal Investigator — Duke University; Joseph P McEvoy, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - John Umstead Hospital, Butner, North Carolina
  - Duke University Medical Center, Durham, North Carolina